CLINICAL TRIAL: NCT03737799
Title: StartRight: Getting the Right Classification and Treatment From Diagnosis in Adults With Diabetes
Acronym: StartRight
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Diabetes UK (Other); University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: CRF243; 203567 (Other: IRAS); CS-2015-15-018 (Other Grant/Funding Number: NIHR); 17/0005624 (Other Grant/Funding Number: Diabetes UK)
Record Dates: First submitted 2018-10-08; First posted 2018-11-13 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; C-peptide; Insulin; Classification
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA, RNA, Cell free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 Age 18-50 at diagnosis: Diagnosed with diabetes within the previous 1 year. Aged between 18 and 50 years at the time of diabetes diagnosis
- Group 2 Late Onset (insulin): Diagnosed with diabetes within the previous 1 year. Aged >50 at the time of diabetes diagnosis and treated with insulin therapy
- Group 3 Late Onset (no insulin): Diagnosed with diabetes within the previous 1 year. Aged >50 at the time of diabetes diagnosis and treated without insulin

SUMMARY:
This study aims to achieve more accurate early classification of diabetes and identification of which patients will rapidly require insulin treatment. The investigators will recruit 1200 participants who have been diagnosed with diabetes in the last year and were aged between 18 and 50 years at the time of diagnosis. The investigators will recruit an additional cohort of 800 participants diagnosed after age 50. The investigators will record clinical features and biomarkers that may help us to determine diabetes type at diagnosis and follow participants for 3 years to assess the development of severe insulin deficiency (measured using C-peptide) and insulin requirement. The investigators will assess utility of clinical features and additional biomarkers in identifying patients with rapid progression to insulin requirement. Findings will be integrated into a freely available clinical prediction models to assist classification of diabetes at diagnosis.

DETAILED DESCRIPTION:
The study is a prospective observational study which will assess the relationship between clinical features and biomarkers at diabetes diagnosis and type of diabetes defined by endogenous insulin secretion at 3 years diabetes duration.

The investigators will recruit a prospective cohort of 1200 adults that have been diagnosed with diabetes within the previous 1 year and aged between 18 and 50 at the time of diagnosis. The investigators will also recruit an additional cohort of 800 participants diagnosed with diabetes in the last year aged >50 at diabetes diagnosis, who will be stratified by insulin treatment (insulin treated n=400).

On recruitment into the study, non-fasting (within 1-5 hours of a meal) blood sample will be collected for baseline analysis biomarker assessment (serum C-peptide, routine biochemistry, Islet autoantibodies (GAD, IA2, ZnT8)) and biobanking. Clinical features will be recorded, including weight, height, waist/hip ratio & blood pressure. Participants will be asked to provide a home post-meal urine sample for Urinary C-Peptide Creatinine Ratio (UCPCR). At 1 year and 2 years post recruitment, participants will be contacted by telephone, email or in person to record concurrent treatment, hypoglycaemia and health service utilisation. Participants will be asked to collect a home post-meal urine sample for Urinary C-Peptide /Creatinine Ratio (UCPCR). HbA1c results will be obtained from participants GP practice or laboratory records.

At the end of the study, 3 years post recruitment, a non-fasting blood sample will be collected for serum C-peptide, routine biochemistry and stored for future biomarker analysis. Weight change, blood pressure, concurrent treatment, hypoglycaemia and health service utilisation data will be also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with diabetes within the previous 12 months.
* Aged ≥18 and ≤50 at the time of diabetes diagnosis* or (additional late onset diabetes cohort) aged >50 at the time of diabetes diagnosis.
* Able and willing to provide informed consent

Exclusion Criteria:

* Gestational diabetes.
* Known secondary diabetes (diabetes considered likely due to medication, cystic fibrosis, pancreatitis, pancreatic cancer, pancreatic surgery, hemochromatosis or Cushing's syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recently diagnosed diabetes patients in primary care, secondary care or community.
Sampling Method: Non-Probability Sample
Enrollment: 1815 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes type defined by insulin requirement at 3 years | 3 years
  Type 1 diabetes = Progression to insulin treatment and severe insulin deficiency (post meal plasma C-peptide <600pmol/L) at 3 years.
  Type 2 diabetes = Lack of requirement for insulin at 3 years (HbA1c <90mmol/mol without insulin treatment or post meal C-peptide ≥ 600pmol/L if insulin treated).

SECONDARY OUTCOMES:
Stimulated plasma C-peptide <200pmol/L at 3 years ('absolute insulin deficiency') | 3 years
  C-peptide <200pmol/L at 3 years = absolute insulin deficiency
C-peptide rate of change (UCPCR and plasma) | 3 years
  The rate of change of UCPCR and plasma C-peptide
Weight change (baseline to 3 years) | 3 years
  Assessment of weight change from baseline to 3 year visit
HbA1c (mean and at 3 years) | 3 years
  Mean HbA1c for all visits and result at 3 years
Self-reported hypoglycaemia & hypoglycaemic awareness (Modified Clark and Gold) | 3 years
  Results from Hypoglycaemia questionnaire
Resilience (CD-RISC questionnaires) | 3 years
  Results from analysis of data from CD-RISC questionnaire
Ketoacidosis (self-reported and confirmed from medical notes) | 3 years
  Self reported Ketoacidosis and confirmation in medical notes
Wellbeing (SF12 questionnaire) | 3 years
  Results from analysis of data from SF12 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Angus G Jones, MBBS MRCP, Principal Investigator — Royal Devon & Exeter NHS Foundation Trust & University of Exeter
Locations (1):
- Anita Hill, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thomas NJ, Lynam AL, Hill AV, Weedon MN, Shields BM, Oram RA, McDonald TJ, Hattersley AT, Jones AG. Type 1 diabetes defined by severe insulin deficiency occurs after 30 years of age and is commonly treated as type 2 diabetes. Diabetologia. 2019 Jul;62(7):1167-1172. doi: 10.1007/s00125-019-4863-8. Epub 2019 Apr 10. PMID 30969375
- [Result] Eason RJ, Thomas NJ, Hill AV, Knight BA, Carr A, Hattersley AT, McDonald TJ, Shields BM, Jones AG; StartRight Study Group. Routine Islet Autoantibody Testing in Clinically Diagnosed Adult-Onset Type 1 Diabetes Can Help Identify Misclassification and the Possibility of Successful Insulin Cessation. Diabetes Care. 2022 Dec 1;45(12):2844-2851. doi: 10.2337/dc22-0623. PMID 36205650
- [Result] Thomas NJ, Hill AV, Dayan CM, Oram RA, McDonald TJ, Shields BM, Jones AG; StartRight Study Group. Age of Diagnosis Does Not Alter the Presentation or Progression of Robustly Defined Adult-Onset Type 1 Diabetes. Diabetes Care. 2023 Jun 1;46(6):1156-1163. doi: 10.2337/dc22-2159. PMID 36802355

DOCUMENTS (1):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03737799/Prot_000.pdf